CLINICAL TRIAL: NCT04939532
Title: SCALE-UP Utah: Community-Academic Partnership to Address COVID-19 Among Utah Community Health Centers
Brief Title: SCALE-UP Utah: Community-Academic Partnership to Address COVID-19 Testing Among Utah Community Health Centers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Association for Utah Community Health (Other); Utah Department of Health (Other); National Institutes of Health (NIH) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, David Wetter, Director, Center for Health Outcomes and Population Equity, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 00136001; 3UL1TR002538-03S2 (NIH)
Record Dates: First submitted 2021-04-07; First posted 2021-06-25 (Actual); Results first posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-12

CONDITIONS: Covid19
Keywords: COVID19; Community Health; Health Information Technology; Population Health; Patient engagement; Rural; Scale up; Screening; Testing; Text messaging; Underserved population; Uninsured; Utah; Uptake
MeSH Terms: conditions — COVID-19; Patient Participation | interventions — Patient Navigation

STUDY DESIGN:
Intervention Model Description: Patient-level, two-arm randomized design for the Population Health Management interventions, TM or TM+PN.
Who Masked: Participant
Masking Description: Patients will not know if they are in the TM or TM+PN intervention arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text-Messaging (TM) (Active Comparator): Population health management intervention that analyzes electronic health record data to automatically identify participants with high risk for either infection or severe disease and proactivity reaches those participants via text message for testing needs (as advised by state and/or federal guidelines) and testing recommendation when applicable. This is a bi-directional text messaging system.
  Interventions: Behavioral: Text-Messaging (TM)
- Text-Messaging plus Patient Navigation (TM+PN) (Active Comparator): Population health management intervention that includes the same bi-directional text-messaging system as Arm 1 (the text messaging condition) with the addition of patient navigation. Patient navigation includes real-time assistance from a community health worker to address barriers, provide motivation, and assist with logistics of COIVD testing.
  Interventions: Behavioral: Text-Messaging (TM); Behavioral: Patient Navigation (PN)

INTERVENTIONS:
Behavioral: Text-Messaging (TM) — Patients in the TM condition will receive HIPAA-compliant bidirectional text messages. Texts will include a brief message regarding COVID-19 risk and will screen the participants for COVID testing needs. Participants who reply "yes" to accepting testing will receive additional messages with a recommendation to be tested, testing locations/hours/phone, and an offer to receive a free at-home test mailed to their home. Patients who reply "no" will receive a text with the clinic phone number and a note to call if anything changes.
Behavioral: Patient Navigation (PN) — Patients in the PN condition, who respond "yes" to accepting testing will receive additional messages with a recommendation to be tested, testing locations/hours/phone, and an offer to receive a free at-home test mailed to their home. In addition they will receive a notice via text message that a Community Health Worker will contact them for patient navigation. At this time, patients will will have the option to opt-out of the phone call from the patient navigator. The Patient Navigation includes advice from navigators to address practical barriers to COVID testing such as logistics, transportation, and expenses as well as behavioral barriers such as hesitancy, fear, and uncertainty.
  Arms: Text-Messaging plus Patient Navigation (TM+PN)

SUMMARY:
SCALE-UP Utah is a community-academic partnership to address COVID-19 among Utah community health centers. The long-term objective of the project is to increase the reach, acceptance, uptake, and long-term sustainability of COVID-19 screening and testing among Utah's Community Health Center patient population. The study will compare two practical, feasible, scalable interventions to increase COVID-19 testing uptake in Utah Community Health Centers:

1. Text Messaging (TM): population health management (PHM) intervention that analyzes EHR data to automatically identify patients with high risk for either infection or severe disease, reaches and screens those patients, and addresses testing logistics using bi-directional text messaging.
2. Patient Navigation (PN): PHM intervention to increase testing uptake among eligible patients (identified via TM) using patient navigation (e.g., motivating patients, addressing logistics and barriers).

The project will employ a rapid cycle research approach in which interventions are tested on a small scale, using short time frames (e.g., <1 month) and cyclical evaluation cycles. This process involves implementing intervention messages with a small number of clinics or patients, evaluating the outcomes, and either adapting the intervention messages based on findings (and retesting) or disseminating effective approaches to additional clinics or patients. A critical feature of these cycles is the ability to quickly test and refine messages in a limited setting before broader implementation. Throughout the study, intervention messages were updated or adapted in response to evolving public health guidelines, testing procedures, and policy recommendations (e.g., priority populations by age group or geographic area, as advised by the Utah Department of Health and Human Services and relevant federal agencies). However, these updates did not alter the fundamental structure of the intervention arms. Participants were randomized to one of two main conditions-Text Messaging (TM) or Text Messaging plus Patient Navigation (TM+PN)-and all participants within a given arm received interventions aligned with their assigned condition. Adaptations occurred within the content and timing of messages or navigation support, but the core components of the interventions remained consistent across participants within each arm. These adaptations were tracked and incorporated into implementation logs but did not constitute distinct intervention arms or conditions.

The specific aims are to:

1. Implement and evaluate PHM interventions for increasing the uptake of COVID-19 testing among CHC patients across Utah. Our primary outcome, Uptake-Eligible, is defined as the proportion of patients who are tested for COVID-19 out of the patients who meet screening criteria for COVID-19 testing. Our study hypothesis is that patients in the TM+PN cohort will have higher rates of uptake-eligible than those in the TM cohort.
2. Examine implementation effectiveness outcomes, as well as characteristics of both clinics and patients that may influence intervention effects and implementation outcomes.

DETAILED DESCRIPTION:
SCALE-UP Utah is a patient-level intervention involving 12 Community Health Centers (39 individual clinics) across Utah. The study is designed to utilize Community Health Center participant records to proactively reach participants for COVID-19 screening and testing. This intervention includes a randomization component between two interventions, text messaging (TM) or text messaging with patient navigation (TM+PN). These two intervention paths are occurring simultaneously within the same clinics.

Text messaging (TM) and text messaging with patient navigation (TM+PN)

Overview:

Participants in the TM condition will receive HIPAA-compliant bidirectional text messages. Texts will include a brief message regarding COVID-19 risk and will screen for if the participant or someone in their close social network should get tested. Participants who reply "yes" will receive additional messages with a recommendation to be tested, testing locations/hours/phone, and an option for an at-home test to be sent directly to their home. Participants who reply "no" will receive a text with the clinic phone number and a note to call if anything changes.

Participants in the TM+PN condition will receive the same text messages as the patients in the TM condition. Text messages will include a brief message regarding risk and will screen for if the patient should get tested. Patients who reply "yes" will receive the same options as those in TM only (a recommendation to be tested, testing locations/hours/phone, and an option for an at-home test to be sent directly to their home) in addition to a notice that a Community Health Worker will contact them for patient navigation. The Patient Navigation includes practical advice from navigators to address barriers to testing such as logistics, transportation, and expenses.

Step One: Primary Data Extraction To identify the cohort for the TM and TM+PN interventions, a subset of EHR data will be manually extracted from the Community Health Centers as text files generated by EHR reports. The first set of EHR reports will contain all patients seen at each of the Community Health Centers in the last 3 years. Subsequent reports will be obtained weekly, including all encounters in the previous week. Data fields will include risk factors such as age, gender, body mass index, encounter diagnoses for medical co-morbidities, participant demographics (e.g., zip code, insurance status, preferred language, race/ethnicity); as well as cellphone number for text messaging and patient navigation.

Step Two: Randomization & Cohort Selection Once the data are securely housed, all participants will be assigned to either the TM or TM+PN arm of the intervention. This assignment will remain consistent throughout the study. Cohort selection will be based on EHR data considering factors such as age, race/ethnicity, language, relevant medical comorbidities, and residence in hotspot areas. These selection criteria are consistent with recommendations from Utah Department of Health and the Centers for Disease Control and Prevention.

Step Three: Implementation SCALE-UP Utah will send HIPPA-compliant bidirectional texts, which is a communication method routinely used by the Community Health Centers, to patients in high risk cohorts. Text messages will be designed by the research team and sent using a HIPPA compliant text messaging service. The text messaging service will retrieve the participant cohort from the study database to send the texts to the participants. The text messages will appear to the participants as having originated from their Community Health Center. As part of their general Community Health Center care, participants have agreed to be contacted by their Community Health Center and text message communication is one of those established contact methods. Text messages will be repeated weekly, as needed, to continuously screen for COVID-19 testing eligibility and to provide updates. Every text message will include the option to reply STOP to opt-out of receiving text messages at any time.

The text messaging and patient navigation arms of the study will proactively provide patients with access to informative resources describing what would happen if they test positive and where to seek help.

ELIGIBILITY:
Inclusion Criteria:

* current patient of a participating community health center
* own a working cellphone,
* have their phone number listed in their existing electronic medical record at a participating clinic,
* speak English or Spanish.

Exclusion Criteria:

* Minors

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44729 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Wetter, MS, PhD, Principal Investigator — University of Utah; Rachel Hess, MD, MS, Principal Investigator — University of Utah; Guilherme Del Fiol, MD, PhD, Principal Investigator — University of Utah
Locations (1):
- Huntsman Cancer Institute/ University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Text-Messaging Plus Patient Navigation (TM+PN): Population health management intervention that includes the same bi-directional text-messaging system as Arm 1 with the addition of patient navigation (PN). PN includes real-time assistance from a community health worker to address barriers, provide motivation, and assist with logistics of COIVD testing.
  Text-Messaging (TM): Patients in the TM condition will receive HIPAA-compliant bidirectional text messages. Texts will include a brief message regarding COVID-19 risk and will screen the participants for COVID testing needs. Participants who reply "yes" to accepting testing will receive messages with a recommendation to be tested, testing locations/hours/phone, and an offer to receive a free at-home test mailed to their home. Patients who reply "no" will receive a text with the clinic phone number.
  PN: Patients in the PN condition, who respond "yes" to accepting testing will receive additional messages with a recommendation to be tested, testing locations/hours/phone, and an offer to receive a free at-home test. In addition they will receive a notice via text message that a Community Health Worker will contact them for patient navigation. At this time, patients will will have the option to opt-out of the phone call from the patient navigator. The Patient Navigation includes advice from navigators to address practical barriers to COVID testing such as logistics, transportation, and expenses as well as behavioral barriers such as hesitancy, fear, and uncertainty.
Period: Overall Study
Arm/Group | Text-Messaging (TM) | Text-Messaging Plus Patient Navigation (TM+PN)
Started | 22145 | 22584
Completed | 22145 | 22584
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Text-Messaging (TM) | Text-Messaging Plus Patient Navigation (TM+PN) | Total
Number analyzed (Participants) | 22145 | 22584 | 44729
Age, Customized [Count of Participants; unit: Participants]
  18-29 years old | 6997 | 6951 | 13948
  30-64 years old | 13354 | 13713 | 27067
  65 and older | 1794 | 1920 | 3714
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 12144 | 12286 | 24430
  Male | 8925 | 9220 | 18145
  Other or unknown | 1076 | 1078 | 2154
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native White | 322 | 355 | 677
  Asian | 197 | 199 | 396
  Black or African American | 286 | 295 | 581
  Native Hawaiian or Pacific Islander | 186 | 199 | 385
  More than one race | 410 | 429 | 839
  Other Race | 2983 | 3088 | 6071
  White | 13975 | 14296 | 28271
  Unknown or Not Reported | 3786 | 3723 | 7509
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10792 | 11135 | 21927
  Not Hispanic or Latino | 9054 | 9198 | 18252
  Unknown or Not Reported | 2299 | 2251 | 4550

OUTCOME MEASURES:

1. Primary Outcome: Reach-TM Engage
Description: Proportion of patients that respond to the Text Messaging intervention.
Time Frame: 12 months
Population: Proportion of patients that respond to the Text Messaging intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Text-Messaging (TM) | Text-Messaging Plus Patient Navigation (TM+PN)
Number analyzed (Participants) | 22145 | 22584
Participants | 2594 | 2401

2. Secondary Outcome: Total Patients Tested for COVID as Indicated in Health Record Out of Total Patient Population in Study. (Uptake-Total)
Description: Proportion of patients tested for COVID-19 out of the total patient population. Confirmation of COVID test as indicated in patient's health record.
Time Frame: 12 months
Population: No participant data were collected or analyzed. Due to rapid changes in testing and eligibility policies, it was not feasible for the state health department and our partnering clinics to track eligibility and collect individualized testing data, as patients may complete their COVID-19 tests at locations that did not share records, or complete a self-test and failed to report the result to the study. Therefore, these outcomes were not measured and will not be collected in the future.
Groups:
- Text-Messaging Plus Patient Navigation (TM+PN): Intervention includes the same bi-directional text-messaging system as Arm 1 (the text messaging condition) with the addition of patient navigation (PN). PN includes real-time assistance from a community health worker (CHW) to address barriers, provide motivation, and assist with logistics of COIVD testing.
  Text-Messaging (TM): See TM arm for details. Patient Navigation (PN): Patients in the PN condition, who respond "yes" to accepting testing will receive additional messages with a test recommendation, testing locations/hours/phone, and an offer to receive a free at-home test mailed to their home. In addition they will receive a notice via text message that a CHW will contact them for patient navigation. At this time, patients will will have the option to opt-out of the phone call from the patient navigator. The PN includes advice from navigators to address practical barriers to COVID testing such as logistics, transportation, and expenses as well as behavioral barriers such as hesitancy, fear, and uncertainty.
Arm/Group | Text-Messaging Plus Patient Navigation (TM+PN) | Text-Messaging (TM)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Reach PN-Engage-Logistics Assistance
Description: Proportion of patients offered Logistics Assistance Patient Navigator (PN-LA) that talk to a PN
Time Frame: 12 months
Population: Proportion of patients offered Logistics Assistance Patient Navigator (PN-LA) that talk to a PN
Measure: Count of Participants; unit: Participants
Arm/Group | Text-Messaging (TM) | Text-Messaging Plus Patient Navigation (TM+PN)
Number analyzed (Participants) | 0 | 470
Participants | 0 | 152

4. Secondary Outcome: Reach PN-Engage-Requested Navigation
Description: Proportion of patients offered Requested Navigation Patient Navigator (PN-RN) that talk to a PN
Time Frame: 12 months
Population: Proportion of patients offered Requested Navigation Patient Navigator (PN-RN) that talk to a PN
Measure: Count of Participants; unit: Participants
Arm/Group | Text-Messaging (TM) | Text-Messaging Plus Patient Navigation (TM+PN)
Number analyzed (Participants) | 0 | 841
Participants | 0 | 56

5. Secondary Outcome: Uptake-Eligible
Description: Proportion of patients tested for COVID-19 out of those who meet screening criteria for testing. For each patient, we will define a separate Uptake-Eligible measurement for each week of the intervention period in which the patient either responds to a text message or contacts his/her Community Health Center to indicate the presence of symptoms or contact with someone with COVID-19 during the current week, but did not do so in the preceding week.
Time Frame: 12 months
Population: as for outcome 2
Groups:
- Text-Messaging Plus Patient Navigation (TM+PN): Population health management intervention that includes the same bi-directional text-messaging system as Arm 1 (the text messaging condition) with the addition of patient navigation. Patient navigation includes real-time assistance from a community health worker to address barriers, provide motivation, and assist with logistics of COIVD testing.
  Text-Messaging (TM): See TM arm for details
  Patient Navigation (PN): Patients in the PN condition, who respond "yes" to accepting testing will receive additional messages with a recommendation to be tested, testing locations/hours/phone, and an offer to receive a free at-home test mailed to their home. In addition they will receive a notice via text message that a Community Health Worker will contact them for patient navigation. At this time, patients will will have the option to opt-out of the phone call from the patient navigator. The Patient Navigation includes advice from navigators to address practical barriers to COVID testing such as logistics, transportation, and expenses as well as behavioral barriers such as hesitancy, fear, and uncertainty.
Arm/Group | Text-Messaging Plus Patient Navigation (TM+PN) | Text-Messaging (TM)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: This project used a non-systematic assessment method to evaluate adverse events. Although adverse events were not routinely assessed, data on adverse events were collected for up to 23 months after a participant's enrollment in the project.
Description: Adapted intervention refers to the adaptation of messages, not interventions. Throughout the study, intervention messages were updated or adapted in response to evolving public health guidelines, testing procedures, and policy recommendations These updates did not alter the fundamental structure of the intervention arms and did not constitute distinct intervention arms or conditions
Arm/Group | Text-Messaging (TM) | Text-Messaging Plus Patient Navigation (TM+PN)
All-Cause Mortality (participants affected / at risk) | 0/22145 | 0/22584
Serious Adverse Events (participants affected / at risk) | 0/22145 | 0/22584
Other Adverse Events (participants affected / at risk) | 0/22145 | 0/22584

LIMITATIONS AND CAVEATS:
The outcomes (Uptake-Eligible) and (Uptake-Total) require the collection of individualized COVID-19 testing data. As COVID testing options evolved throughout the pandemic, our ability to track eligibility and collect testing outcomes from all available sources greatly diminished. We have no individualized testing data and therefore are unable to analyze Uptake-Total and Uptake-Eligible outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2022-02-23): https://cdn.clinicaltrials.gov/large-docs/32/NCT04939532/Prot_000.pdf